





Please <u>initial</u>

box. <u>Do</u> not tick

## CONSENT FORM

Plasma biomarkers in stratifying patients referred via the lower gastro-intestinal (LGI) suspected cancer two-week wait (2WW) pathway MOTION study

Participant ID:

| Please read the statements below. Put <u>initials</u> of your name in the boxes if you agree, put an X in any box where you do not agree and sign the form. <b>Use BLACK pen only</b> |
|---|
| 1. I confirm that I have read and understand the Patient Information Sheet dated [DATE] (version |
| [VERSION NUMBER]) for MOTION study. I have had the opportunity to consider the information, ask |
| questions and have had these answered satisfactorily. |
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without |
| giving any reason and without my care or legal rights being affected. |
| 3. I agree that confidential study data collected prior to my withdrawal from the MOTION study can be |
| used in the study reports. I understand that if I lose capacity to consent during the study I will be |
| withdrawn and the agreed data already collected can be used. |
| 4. I understand that relevant sections of my medical notes and data collected during the MOTION study |
| may be looked at by individuals from the Queen Mary, University of London (QMUL) or Barts Health |
| NHS Trust (BHT). I give permission for these individuals to have access to my records. |
| 5. I agree for my contact details and identifiable personal data to remain within the study site (QMUL or |
| BHT). I understand that coded personal data, including data from medical records and study-specific |
| data, may be shared with collaborators within the EU for the purposes of research and data analysis. |
| 6. I agree to my GP or/ and referring doctors being informed of my participation in the MOTION study. |
| 7. I understand that the study data collected will be used for medical research only. I will be given a |
| Unique Identification Number (UIN/ Patient ID) in order to ensure that my data is confidential and will not |
| directly identify me. |
| 8. I agree my confidential study data can be used in the analysis and reporting of the study findings. |
| 9. I understand that participants will be asked to give a 20 millilitres of blood sample, to be taken in clinic |
| or in endoscopy or in the radiology department. I consent to having my blood drawn. |
| 10. I understand that a laboratory will analyse my blood sample and the MOTION study team will record |
| this information. |
| 11. I understand that a part of my blood sample will be transported to our collaborators in France. |
| A portion of the blood sample collected for this study will be sent to Progastrin Manufacturing, Biodena |

Care, located at Cap Sigma-Zac Euromedicine II, 1682 Rue de la Vasière, 34790 Grabels, France, for

12. I understand that this MOTION study also involves the analysis of my DNA and RNA from plasma

13. I understand that the storage of my samples will be pseudonymised (labelled with an ID number

instead of personally identifying information) and outcomes of the analysis are unlikely

Copies: 1 for patient; 1 for study team, 1 for medical notes IRAS number: 321809 Patient Informed Consent Form\_v1.5\_7th April 25

the purpose of biomarker analysis.

and I agree for genetic analysis to be done.







| to have any implications for me personally. | | | |
|---|---|---|---|
| 14. I understand that my contact details will be kept in order for the study team to communicate with me | | | |
| about the study and for QMUL to retain study-related information for 5 years after the study ends, after | | | |
| which point all study materials will be destroyed. | | | |
| 15. I understand that relevant sections of my medical notes and data collected during | | | |
| the study may be looked at by individuals from QMUL or BHT, from regulatory authorities or | | | |
| from the NHS Trust, where it is relevant to my taking part in this research. I give permission for | | | |
| these individuals to have access to my records. | | | |
| 16. I agree to take part in the study. | | | |
| 17. OPTIONAL | | | |
| I agree to be contacted by the study team to complete a survey at the end of the two-week wait | | | |
| pathway using my contact details. | | | |
| 18. OPTIONAL | | | |
| I prefer to be informed and receive information about this questionnaire through the following | | | |
| methods. | □ phone intervie | w 🗆 SMS | |
| 19. OPTIONAL | | | |
| I understand that the information collected about me will be used to support other research in the | | | |
| future and may be shared anonymously with other researchers. | | | |
| 20. OPTIONAL | | | |
| Following the present study, any residual (left-over) plasma may be stored and used by the research | | | |
| team at QMUL, for future research studies. Any future studies will have Ethics Committee permission. | | | |
| 21. OPTIONAL | | | |
| I agree to be contacted about future related stud | lies. | | |
| Print Name of Participant: | Date: | Participant's Signature: | |
| Print Name of person taking consent: | Date: | Signature of person taking cor | nsent: |